CLINICAL TRIAL: NCT01832857
Title: An Open Label, Phase 2 Trial to Evaluate the Safety, Tolerability and Efficacy of CPI-613 in Cancer Patients
Brief Title: Phase 2 Safety, Tolerability and Efficacy Study of CPI-613 in Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-CPI-613-023
Record Dates: First submitted 2013-04-12; First posted 2013-04-16 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Cancer
Keywords: metastatic; advanced; solid tumor; cancer; colon cancer; hepatocellular carcinoma; breast cancer; lung cancer; gastric cancer; esophageal cancer
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Carcinoma, Hepatocellular; Breast Neoplasms; Lung Neoplasms; Stomach Neoplasms; Esophageal Neoplasms | interventions — devimistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPI-613 Alone (Experimental): This arm is for patients that have failed, or are not eligible for, all available therapies. CPI-613 drug product, provided in concentrated form at 50 mg/mL, must be diluted with D5W prior to administration. CPI-613 is to be infused intravenously (IV) via a central venous catheter. CPI-613 will be given 2x weekly, administered on Days 1 and 4 of each of the 3 treatment weeks, followed by a week of rest. The dose of CPI-613 will be 3,000 mg/m2 infused IV over 2 hours (this is the maximum tolerated dosing [MTD]), via a central venous catheter with D5W running at a rate of about 125-150 mL/hr.
  Interventions: Drug: CPI-613

INTERVENTIONS:
Drug: CPI-613 — CPI-613 drug product, provided in concentrated form at 50 mg/mL, must be diluted with D5W prior to administration. CPI-613 is to be infused intravenously (IV) via a central venous catheter. CPI-613 will be given 2x weekly, administered on Days 1 and 4 of each of the 3 treatment weeks, followed by a week of rest. The dose of CPI-613 will be 3,000 mg/m2 infused IV over 2 hours (this is the maximum tolerated dosing [MTD]), via a central venous catheter with D5W running at a rate of about 125-150 mL/hr.
  Other Names: 6,8-bis-benzylsulfanyloctanoic acid; 6,8-bis(benzylthio)octanoic acid; 6,8-bis-benzylsulfonyloctanoic acid; Bylantra (tentative)

SUMMARY:
This Phase II study is conducted to assess the safety and efficacy of CPI-613 in patients with advanced and/or metastatic solid tumors for whom there there is no available therapy to provide clinical benefit or for those who have refused further standard therapy. The primary outcome measure is Overall Survival (OS). The secondary outcome measures are: Response Rate (RR), Progression-Free Survival (PFS), and safety.

DETAILED DESCRIPTION:
Open-Label Single-Arm Design: This is an open-label study, and investigators and subjects are not blinded to the treatment. Also, the assignment of patients will not be randomized, since this is a single-arm study.

Treatment with CPI-613: A treatment cycle is 4 weeks, with CPI-613 given on Days 1 and 4 of the first 3 weeks.

Dose and Sample Size: The dose of CPI-613 is 3,000 mg/m2. This is Maximum Tolerated Dose (MTD) determined from the Phase I dose-escalated trial, Study# CL-CPI-613-009 (conducted in patients with hematologic malignancies under IND 107,800). This dose has also been found to be well tolerated in another Phase I dose-escalated trial, Study# CL-CPI-613-002 (conducted in patients with solid tumor under IND 74,530). There will be 20 evaluable patients with each tumor type. Once there are 20 evaluable patients with a particular tumor type has been treated with at least 1 cycle, no patients of the same tumor type will be accrued. Dosing Delay and Dose Modification of CPI-613 in the Event of Adverse Events: For adverse events unrelated to serum creatinine elevation or reduction in renal function but are possibly related to CPI-613, the occurrence of Grade 1 toxicity does not generally require dose modification for subsequent doses for that patient. However, if Grade 2 toxicity (other than alopecia and nausea) probably related to CPI-613 develops, treatment is to be withheld and can resume only after the Grade 2 toxicity has been reduced to Grade 1 or below, and the dose level for subsequent doses for that patient will be reduced by 25% of the dose at which such Grade 2 toxicity occurs. Grade 2 alopecia and nausea do not require withholding treatment or dose reduction. If Grade 3 or 4 toxicity probably related to CPI-613 develops, dosing of CPI-613 of that patient will be withheld and the patient shall be monitored for recovery from, and reversibility of, such Grade 3 or 4 toxicity. To resume treatment with CPI-613 for a patient who has had CPI-613-related Grade 3 or 4 toxicity, the Grade 3 or 4 toxicity must be reduced to Grade 1 or below, and the dose level for subsequent doses for that patient will be reduced to 50% of the dose at which such Grade 3 or 4 toxicity occurs.

For adverse events related to creatinine elevation or reduction in renal function that are possibly related to CPI-613, dosing of the patient will be withheld even if the severity level is Grade 1 or above. Treatment can resume only after the toxicity has been reduced to Grade 0. The dose level for subsequent doses for that patient will be reduced by 15% if the severity level is of Grade 1, by 25% for Grade 2 toxicity, and by 50% for Grade 3 or 4 toxicity.

Furthermore, if the toxicity possibly related to CPI-613 is acute renal failure and the severity level is Grade 3 or 4, further patient enrollment will be temporarily suspended in order to enable assessment of the following aspects of the trial and implementation of corrective measures or protocol amendment, and if necessary:

* compliance of the study sites and investigators to the study protocol
* evaluation of the appropriateness of the procedures for monitoring renal function

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced and/or metastatic, histologically or cytologically documented solid tumors, for whom there is no available therapy shown to provide clinical benefit or for those who have refused further standard therapy
* Eastern Cooperative Oncology Group (ECOG) performance status being 0-2
* Expected survival >3 months
* 18 years of age or older of both genders
* Women of child-bearing potential must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation.
* Fertile men must practice effective contraceptive methods during the study, unless documentation of infertility exists
* Mentally competent, with an ability to understand and willingness to sign the informed consent form
* No radiotherapy, treatment with cytotoxic agents (except CPI-613), or treatment with biologic agents within 3 weeks prior to treatment with CPI-613. At least 2 weeks must have elapsed from any prior surgery or hormonal therapy. Patients must have fully recovered from the acute toxicities of any prior treatment with any anti-cancer drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment). Patients with persisting, stable chronic toxicities from prior treatment ≤Grade 1 are eligible, but must be documented as such.
* Laboratory values ≤2 weeks must be:
* Adequate hematologic (white blood cell [WBC] ≥3500 cells/mm3 or ≥3.5 bil/L; platelet count ≥150,000 cells/mm3 or ≥150 bil/L; absolute neutrophil count [ANC] ≥1500 cells/mm3 or ≥1.5 bil/L; and hemoglobin (Hgb) ≥9 g/dL or ≥90 g/L).
* Adequate hepatic function (aspartate aminotransferase [AST/SGOT] ≤3x upper normal limit [UNL], alanine aminotransferase [ALT/SGPT] ≤3x UNL (≤5x UNL if liver metastases present), bilirubin ≤1.5x UNL).
* Adequate renal function (serum creatinine ≤2.0 mg/dL or 177 μmol/L, and blood urea nitrogen [BUN] ≤25 mg/dL).
* Adequate coagulation ("International Normalized Ratio or INR must be ≤1.5")

Exclusion Criteria:

* Serious medical illness
* Any active uncontrolled bleeding or patients with a bleeding diathesis
* Patients with active central nervous system (CNS) or epidural tumor
* Pregnant women, or women of child-bearing potential not using reliable means of contraception
* Lactating females
* Fertile men unwilling to practice contraceptive methods during the study period
* Life expectancy less than 3 months
* Unwilling or unable to follow protocol requirements
* Dyspnea with minimal to moderate exertion, or patients with pleural, pericardial, or peritoneal effusions
* Active heart disease including but not limited to symptomatic congestive heart failure, symptomatic coronary artery disease, symptomatic angina pectoris, symptomatic myocardial infarction, arrhythmias requiring medication, or symptomatic congestive heart failure.
* A marked baseline prolongation of QT/QTc interval; a history of additional risk factors for torsade de pointes.
* Requirement for immediate palliative treatment of any kind including surgery
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients
* Albumin <2.5 g/dL or <25 g/L
* Evidence of active infection, or serious infection, with the past month
* Patients with known HIV infection.
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 3 weeks prior to initiation of CPI-613 treatment.
* Patients who have received immunotherapy of any type within the past 4 weeks prior to initiation of CPI-613 treatment
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months
* Troponin I above institution limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Monitored until participants pass away, for an expected average of 6 months.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Monitored during treatment with CPI-613 and until participants passed away, which will be an expected average of 6 months.
Safety | Monitored just before study treatment, and during study treatment at the end of every 4-week treatment cycle, for an expected average of 20 weeks.
  Safety assessment will be based on clinical signs, vital signs, blood work, adverse events (AEs), serious adverse events (SAEs), etc.
Response Rate | Monitored at the end of every 4-week treatment cycle during treatment with CPI-613, for an expected average of 20 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: King C Lee, Ph.D., Study Chair — Cornerstone Pharmaceuticals
Locations (1):
- Eastchester Center for Cancer Care, The Bronx, New York, United States

REFERENCES:
- [Derived] Liu N, Yan M, Tao Q, Wu J, Chen J, Chen X, Peng C. Inhibition of TCA cycle improves the anti-PD-1 immunotherapy efficacy in melanoma cells via ATF3-mediated PD-L1 expression and glycolysis. J Immunother Cancer. 2023 Sep;11(9):e007146. doi: 10.1136/jitc-2023-007146. PMID 37678921